CLINICAL TRIAL: NCT02152579
Title: Open Monocentric Clinical Study for the Evaluation of Efficacy and Safety of 20 mg Monocordil Tablets Manufactured by Laboratórios Baldacci in Patients With Stable Angina
Brief Title: Efficacy and Safety of Monocordil Manufactured by Laboratórios Baldacci
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratórios Baldacci S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATC 001/14
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Stable Angina
Keywords: Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isosorbide-5-mononitrate, tablet (Experimental): Single treatment arm.
  Interventions: Drug: Isosorbide-5-mononitrate

INTERVENTIONS:
Drug: Isosorbide-5-mononitrate — Patients will receive 20mg monocordil tablets (Baldacci Laboratories).
  Other Names: Monocordil

SUMMARY:
Phase III clinical study for the evaluation of clinic and cardiologic effects of isosorbide mononitrate from the incidence of events (angina episodes).

This is an open, comparative, monocentric trial. The hypothesis, regarding the number of angina episodes, to be tested are:

* H0: μD = 0 ot H0: μAfter = μBefore
* HA: μD ≠ 0 ot HA: μBefore ≠ μAfter

DETAILED DESCRIPTION:
Phase III study, monocentric, open, with a single treatment arm in patients with stable angina to evaluates efficacy and safety. The study will be sponsored by pelo Laboratórios Baldacci. All patients who participate in the study shall sign two copies of the informed consent form. The inclusion of patients is expected to last until 12 months from the approval of the Ethics Committee and ANVISA.

Follow up will last at least 2 weeks for each included patient. A total of 86 patients will be recruited for this study and all of them will initiate treatment with 20 mg monocordil tablets. After 2 consecutive weeks using the investigational product (+2 days), the patients will be evaluated again, particularly for the parameters under study, this is, quantity and severity of angina episodes and adverse events. The selected patients shall also be 18-80 years old of both genders, with proved diagnosis of stable angina through clinical exams such as ECG, physical effort tests or similar. Patients will receive 20mg monocordil tablets (Baldacci Laboratories).

The evaluations will take place in two opportunities: one at the visit of medical evaluation and recruitment in the study (along with the deliver of the study medication and a diary) and the second one after 2 weeks (+2 days) of use of 20mg monocordil tablets for medical evaluation and discharge of the study (return of the diary and medication accountability).

ELIGIBILITY:
Inclusion Criteria:

* Capacity for understanding and agreement in signing the informed consent form
* Age 18 between 18 and 80 years old
* Have a diagnosis of stable angina, proved by ECG, test of physical effort or similar
* Not being under treatment with other nitrate for stable angina
* Medical indication for the use of isosorbide mononitrate (Monocordil)

Exclusion Criteria:

* Presence or serious comorbidities (under judgement of the investigator)
* Allergy to any of the component of the investigational product
* Pregnant female patients, brest feeding and/or in fertile condition who wish to get pregnant during the study and deny the use of contraceptives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Absolute number of episodes of angina | 15 days
  The absolute parameter of incidence of improvement will be used as primary endpoint, being considered as improvement the reduction in the number of events in 15 days, after the beginning of the intake of the study medication, and the intensity of the angina crisis

SECONDARY OUTCOMES:
Adverse events | 15 days
  The secondary endpoints to be used are the other parameters supplied by the diary (incidence and intensity of Adverse Events).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo G Modolo, MD, Principal Investigator — ATCGen
Locations (1):
- Clinicordis, Campinas, São Paulo, Brazil